CLINICAL TRIAL: NCT03674970
Title: Effects of Random Nicotine Delivery on Smoking Cessation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Patricia Sue Grigson, Director, Penn State Addiction Center for Translation and Professor of Neural and Behavioral Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9977; R21DA038775 (NIH)
Record Dates: First submitted 2018-09-14; First posted 2018-09-18 (Actual); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Smoking Cessation; Cigarette Smoking; Smoking (Tobacco) Addiction
Keywords: smoking cessation; nicotine film; nicotine delivery; random nicotine delivery
MeSH Terms: conditions — Smoking Cessation; Cigarette Smoking; Smoking; Behavior, Addictive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Random Nicotine Delivery (Experimental): One 0 mg or 4 mg nicotine film every 3-4 hours for a total of four films per day (not to exceed three non-consecutive 4 mg films in one day) for 6 weeks.
  Interventions: Drug: Nicotine Film
- Steady State Nicotine Delivery (Active Comparator): One 2 mg nicotine film every 3-4 hours for a total of four films per day for 6 weeks.
  Interventions: Drug: Nicotine Film
- Placebo Control (Placebo Comparator): One 0 mg nicotine film every 3-4 hours for a total of four films per day for 6 weeks.
  Interventions: Drug: Nicotine Film

INTERVENTIONS:
Drug: Nicotine Film — Three doses of nicotine films will be used in this project: 0 mg, 2 mg, and 4 mg.
  The active pharmaceutical ingredient in the nicotine film product is nicotine polacrilex (20%, USP). The film has a muco-adhesive property and allows nicotine to be absorbed through the oral mucosa. After placement in the oral cavity, the nicotine film dissolves in less than five minutes. The film is in the form of 1 inch x 1 inch square and weighs about 100 mg. Nicotine films are not available in the United States in a non-investigational setting.

SUMMARY:
The objective of this study is to determine whether treatment with random nicotine delivery via a nicotine film both before and after the target quit date will facilitate smoking cessation relative to treatment with steady state delivery or placebo.

The investigators hypothesize that smoking cessation will be greater in subjects assigned to a random nicotine delivery regimen (as compared to those assigned to a steady state or placebo regimen). The nicotine film product is not part of the standard of care and is not available in non-investigational settings in the United States.

DETAILED DESCRIPTION:
This project is a prospective parallel-group, randomized, double-blind, placebo-controlled study in which 45 current cigarette smokers who are interested in quitting will be randomly allocated to one of three possible nicotine film treatment regimens:

1. Random nicotine delivery (a combination of four 0 mg and 4 mg films daily not to exceed three non-consecutive 4 mg films in one day and to maintain an average of 8 mg of nicotine per day through 7 days for 6 weeks total).
2. Steady state nicotine delivery (2, 2, 2, 2 mg films daily for 6 weeks total)
3. Placebo delivery (0, 0, 0, 0 mg films daily for 6 weeks total)

Prior to assignment in one of the above treatment groups, all participants will take part in a 1-week baseline period to assess normal smoking behavior and nicotine dependence. Following randomization to their assigned treatment group at Visit 2, participants will be instructed to smoke cigarettes as they feel necessary over the next two weeks while using the nicotine films as directed (i.e., one film every 3-4 hours for a total of four films per day). After two weeks of pre-cessation treatment, participants will be asked completely cease cigarette smoking and to only use their assigned nicotine films as directed. Participants will be supported in their quitting efforts with regular contacts both in person at the Penn State Milton S. Hershey Medical Center and over the phone.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-55
* Smoke ≥10 cigarettes/day for at least the past 12 months
* Exhaled CO measurement ≥6 ppm at baseline visit
* Interested in completely ceasing cigarette consumption and using a nicotine film product as directed
* Willing to attend regular visits over a 6-week period (not planning to move, not planning extended vacation, no planned surgeries)
* Able to read and write in English
* Able to understand and consent to study procedures

Exclusion Criteria:

* Unstable or significant medical conditions and conditions such as elevated blood pressure (systolic >159 mmHg or diastolic >99mmHg at baseline), COPD, and those conditions that are likely to affect biomarker data such as kidney or liver disease
* Individuals with sodium-restricted diet, heart disease, recent heart attack, irregular heartbeat, stomach ulcers, or diabetes as well as those taking prescription medications for depression or asthma as indicated under "Warnings" section on FDA approved NRT Drug Facts Label
* More than weekly use in the past 3 months of illegal drugs or prescription drugs that are not being used for medically prescribed purposes
* Use of non-cigarette nicotine delivery product in the prior 7 days (including cigars, pipes, chew, snus, hookah, electronic cigarette and marijuana mixed with tobacco)
* Use of an FDA approved cessation medication in the past 7 days (any NRT, Chantix, Wellbutrin)
* Women who are pregnant (verified by urine pregnancy test at baseline visit), trying to become pregnant, or nursing
* Uncontrolled mental illness or substance abuse or inpatient treatment for these conditions in the past 6 months
* Any previous adverse reaction to NRT
* Any other condition, serious illness, or situation that would, in the investigator's opinion, make it unlikely that the participant could comply with the study protocol
* Other member of household currently participating in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia S Grigson, PhD, Principal Investigator — Penn State College of Medicine; Jonathan Foulds, PhD, Principal Investigator — Penn State College of Medicine; Christopher Sciamanna, MD, Study Director — Penn State College of Medicine
Locations (1):
- Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Random Nicotine Delivery: One 0 mg or 4 mg nicotine film every 3-4 hours for a total of four films per day (not to exceed three non-consecutive 4 mg films in one day) for 6 weeks.
  Nicotine Film: Three doses of nicotine films will be used in this project: 0 mg, 2 mg, and 4 mg.
  The active pharmaceutical ingredient in the nicotine film product is nicotine polacrilex (20%, USP). The film has a muco-adhesive property and allows nicotine to be absorbed through the oral mucosa. After placement in the oral cavity, the nicotine film dissolves in less than five minutes. The film is in the form of 1 inch x 1 inch square and weighs about 100 mg. Nicotine films are not available in the United States in a non-investigational setting.
- Steady State Nicotine Delivery: One 2 mg nicotine film every 3-4 hours for a total of four films per day for 6 weeks.
  Nicotine Film: Three doses of nicotine films will be used in this project: 0 mg, 2 mg, and 4 mg.
  The active pharmaceutical ingredient in the nicotine film product is nicotine polacrilex (20%, USP). The film has a muco-adhesive property and allows nicotine to be absorbed through the oral mucosa. After placement in the oral cavity, the nicotine film dissolves in less than five minutes. The film is in the form of 1 inch x 1 inch square and weighs about 100 mg. Nicotine films are not available in the United States in a non-investigational setting.
- Placebo Control: One 0 mg nicotine film every 3-4 hours for a total of four films per day for 6 weeks.
  Nicotine Film: Three doses of nicotine films will be used in this project: 0 mg, 2 mg, and 4 mg.
  The active pharmaceutical ingredient in the nicotine film product is nicotine polacrilex (20%, USP). The film has a muco-adhesive property and allows nicotine to be absorbed through the oral mucosa. After placement in the oral cavity, the nicotine film dissolves in less than five minutes. The film is in the form of 1 inch x 1 inch square and weighs about 100 mg. Nicotine films are not available in the United States in a non-investigational setting.
Period: Overall Study
Arm/Group | Random Nicotine Delivery | Steady State Nicotine Delivery | Placebo Control
Started | 15 | 15 | 15
Completed | 12 | 8 | 12
Not Completed | 3 | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Random Nicotine Delivery | Steady State Nicotine Delivery | Placebo Control | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (9.2) | 44.0 (8.1) | 43.2 (5.8) | 43.1 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 11 | 34
  Male | 5 | 2 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 15 | 14 | 15 | 44
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 14 | 15 | 13 | 42
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 15 | 45
Cigarettes Per Day [Mean (Standard Deviation); unit: Cigarettes per day] | 19.6 (7.7) | 18.8 (6.6) | 16.8 (4.5) | 18.4 (6.4)
Fagerstrom Test for Nicotine Dependence Total Score [Mean (Standard Deviation); unit: Scores on a scale] — The Fagerstrom Test for Nicotine Dependence is a 6 item questionnaire to assess dependence on cigarettes. The total score is a sum of each item's score. The range of the total score is 1-10. Scores indicate the following: 1-2 = very low dependence; 3-4 = low dependence; 5 = moderate dependence; 6-7 = high dependence; 8+ = very high dependence.
  Scores on a scale | 5.0 (1.4) | 4.9 (1.1) | 4.3 (1.8) | 4.7 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Cigarettes Smoked Per Day (CPD)
Description: CPD is measured with the use of daily cigarette logs which are completed daily by participants and returned to the study center at each visit. The CPD measure will be the average of the past 7 days.
Time Frame: Baseline and 4 weeks after Target Quit Date
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Random Nicotine Delivery | Steady State Nicotine Delivery | Placebo Control
Number analyzed (Participants) | 15 | 15 | 15
cigarettes per day | -10.3 (6.1) | -9.0 (8.0) | -7.6 (5.3)
Statistical Analysis 1: Comparison: Random Nicotine Delivery vs Steady State Nicotine Delivery vs Placebo Control; Test type: Other; p = .55, ANOVA

2. Primary Outcome: Change in Exhaled Carbon Monoxide (CO) Measurement
Description: Mean change in exhaled CO (parts per million [ppm])
Time Frame: Baseline and 4 weeks after Target Quit Date
Measure: Mean (Standard Deviation); unit: parts per million
Arm/Group | Random Nicotine Delivery | Steady State Nicotine Delivery | Placebo Control
Number analyzed (Participants) | 15 | 15 | 15
parts per million | -16 (18.6) | -5.9 (13.4) | -10.5 (9.1)
Statistical Analysis 1: Comparison: Random Nicotine Delivery vs Steady State Nicotine Delivery vs Placebo Control; Test type: Other; p = .2146, ANOVA

3. Secondary Outcome: Change in Questionnaire of Smoking Urges-Brief (QSU-Brief) Total Score
Description: The QSU-Brief, with a possible total score range of 10 to 70, is an instrument used to measure cigarette craving. A score of 10 on this scale indicates very low cigarette craving, while a score of 70 indicates very high cigarette craving.
Time Frame: Baseline and 4 weeks after Target Quit Date
Measure: Mean (Standard Deviation); unit: QSU Total Score
Arm/Group | Random Nicotine Delivery | Steady State Nicotine Delivery | Placebo Control
Number analyzed (Participants) | 15 | 15 | 15
QSU Total Score | -.55 (1.46) | -.55 (1.36) | -.11 (.97)
Statistical Analysis 1: Comparison: Random Nicotine Delivery vs Steady State Nicotine Delivery vs Placebo Control; Test type: Other; p = .5642, ANOVA

4. Secondary Outcome: Change in Fagerstrom Test for Nicotine Dependence (FTND) Total Score
Description: Nicotine dependence will be assessed via the FTND, a measure with total scores ranging from 0 (very low dependence) to 10 (very high dependence).
Time Frame: Baseline and 4 weeks after Target Quit Date
Measure: Mean (Standard Deviation); unit: FTND Total Score
Arm/Group | Random Nicotine Delivery | Steady State Nicotine Delivery | Placebo Control
Number analyzed (Participants) | 15 | 15 | 15
FTND Total Score | -1.1 (1.44) | -.53 (.92) | -.53 (1.46)
Statistical Analysis 1: Comparison: Random Nicotine Delivery vs Steady State Nicotine Delivery vs Placebo Control; Test type: Other; p = .4353, ANOVA

5. Secondary Outcome: Subjective Ratings Scale for Nicotine Film Use
Description: The scale is comprised of 21 items. Each item is rated on a scale 1-7, where 1 is equal to not at all and 7 is equal to extremely. The total score is the average score of all 21 items. The total score ranges from 1-7.
Time Frame: 4 weeks after Target Quit Date
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Random Nicotine Delivery | Steady State Nicotine Delivery | Placebo Control
Number analyzed (Participants) | 13 | 11 | 15
score on a scale | 3.32 (.71) | 2.82 (.46) | 2.74 (.57)
Statistical Analysis 1: Comparison: Random Nicotine Delivery vs Steady State Nicotine Delivery vs Placebo Control; Test type: Other; p = .0348, ANOVA

6. Secondary Outcome: Side Effects From Nicotine Film Use
Description: Total score ranges from 0 - 36 with lower scores indicating lesser side effects.
Time Frame: 4 weeks after Target Quit Date
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Random Nicotine Delivery | Steady State Nicotine Delivery | Placebo Control
Number analyzed (Participants) | 13 | 11 | 15
score on a scale | 17.77 (4.32) | 15.36 (3.32) | 17.13 (5.15)
Statistical Analysis 1: Comparison: Random Nicotine Delivery vs Steady State Nicotine Delivery vs Placebo Control; Test type: Other; p = .4040, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at each follow-up visit over a period of 7 weeks total.
Arm/Group | Random Nicotine Delivery | Steady State Nicotine Delivery | Placebo Control
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 9/15 | 11/15 | 8/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Random Nicotine Delivery (N=15) | Steady State Nicotine Delivery (N=15) | Placebo Control (N=15)
Dyspepsia (Gastrointestinal disorders) | 4 | 2 | 1
Hiccups (Gastrointestinal disorders) | 2 | 5 | 0
Vomitting (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 4
Anxiety (Psychiatric disorders) | 1 | 1 | 0
Other (Investigations) | 0 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/70/NCT03674970/Prot_SAP_000.pdf